CLINICAL TRIAL: NCT02875652
Title: Study of Circulating Tumoral DNA Evolution in Plasma in Choroidal Melanoma
Brief Title: Circulating Tumoral DNA in Choroidal Melanoma (ctDNA MU)
Acronym: ctDNA MU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2012-08
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Choroidal Melanoma
Keywords: circulation tumor DNA; choroidal melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sampling (Experimental)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — 3 vials of 7,5 ml of peripherical blood will be collected at each blood sample.

SUMMARY:
Quantification and follow-up during 3 years of circulating tumoral DNA in patients with choroidal melanoma

DETAILED DESCRIPTION:
This study is a prospective, open-labelled, monocentric trial. The aim is to observe, in patient with choroidal melanoma (any stage of the disease), the prevalence of the circulating tumor DNA at the diagnostic and its evolution during 3 years.

The patient will have a blood sample at the following times :

* T0: before treatment of the primary tumor.
* T1: 1 months after the end of the local treatment.
* T2: at 7 months.
* Tn: every 6 months up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or more.
* Patient with a recent choroidal melanoma before the start of the specific treatment.
* Patient able to stand a blood collection.
* Work-up for extension (CT).
* Patient explanation given and consent information signed or by legal representative

Exclusion Criteria:

* Patient without social protection / insurance.
* Person deprived of liberty or under guardianship.
* Inability to submit to medical monitoring of the trial for reasons of geography, social or psychological

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2013-03-21 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Assesment of the change of the circulating tumor DNA from baseline at 3 years | T0: before treatment; T1: 1 month after local treatment; T2: at 7 months; Tn : every 6 months up to 3 years.

SECONDARY OUTCOMES:
Compare the treatment effects of the primary tumor (protontherapy, iodine plaque, enucleation) on the rate of circulating tumoral DNA. | 3 years
Comparison of the circulating tumor DNA rate to hepatic imaging if available. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Desjardins, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).